CLINICAL TRIAL: NCT01783990
Title: Pediatric Hydroxyurea Phase III Clinical Trial (BABY HUG) Follow-up Observational Study II Protocol
Acronym: BABY HUG
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: HHSN268201200023C
Record Dates: First submitted 2013-02-01; First posted 2013-02-05 (Estimated); Results first posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2016-09

CONDITIONS: Sickle Cell Anemia
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hydroxyurea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stored blood and urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Active: Complete blood counts (CBCs), reticulocytes, differential, lactate dehydrogenase (LDH), bilirubin and alanine transaminases (ALTs), cystatin C, blood urea nitrogen (BUN), Creatinine, fetal hemoglobin (HbF), pit counts, Howell Jolly Body (HJB), and urine microalbumin:creatinine ratio were collected at study entry, annually, and exit to Follow-Up Study II. Variable-diversity-joining (VDJ) and a stored blood sample were collected at study entry and study exit. Additional tests that include liver/spleen scan, abdominal sonogram, pulmonary function testing, magnetic resonance imaging (MRI) / magnetic resonance angiography (MRA), cardiac echocardiogram, or neuropsychology testing were collected once during the study when the child was 10 years old.
  Interventions: Drug: Hydroxyurea
- Passive: Complete blood counts (CBCs), reticulocytes, differential, lactate dehydrogenase (LDH), bilirubin and alanine transaminases (ALTs), cystatin C, blood urea nitrogen (BUN), Creatinine, fetal hemoglobin (HbF), pit counts, Howell Jolly Body (HJB), variable-diversity-joining (VDJ), urine microalbumin:creatinine ratio and a stored blood sample were collected at study entry and exit to Follow-Up Study II. Additional tests that include liver/spleen scan, abdominal sonogram, pulmonary function testing, MRI/MRA, cardiac echocardiogram, or neuropsychology testing were collected as part of clinical care.
  Interventions: Drug: Hydroxyurea

INTERVENTIONS:
Drug: Hydroxyurea — Parents and child's doctor may plan to use or not to use hydroxyurea.

SUMMARY:
The BABY HUG Treatment Study was designed to see if treatment with the drug hydroxyurea (also called HU) in children with sickle cell disease could prevent organ damage, especially in the spleen and kidneys. There was also a chance that treatment could prevent painful crises, lung disease, stroke, and blood infection.

DETAILED DESCRIPTION:
The current observational trial, Follow-Up Study ((FUS) II includes enhanced neuropsychological, brain, cardiac, and pulmonary evaluations for this very well characterized cohort of subjects. Measures of spleen and renal function and markers of DNA damage will continue to be collected. Assessment of other target organs in sickle cell disease including pulmonary and cardiac function will be performed in addition to evaluation of developmental aspects of sickle cell disease (SCD) and potential HU toxicity.

ELIGIBILITY:
Inclusion Criteria:

* All subjects enrolled in the BABY HUG Follow-Up I Study who participated for at least 24 months are eligible for the Follow-Up Study II

Exclusion Criteria:

* Subjects that have received a Stem Cell Transplant are not eligible for enrollment

Ages: 24 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All subjects enrolled in the BABY HUG Follow-Up I Study who participated for at least 24 months are eligible for the Follow-Up Study II.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2012-10; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Assmann, PhD, Principal Investigator — New England Research Institutes, Watertown, MA
Locations (14):
- United States (14):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Children's National Medical Center Center for Cancer and Blood Disorders, Washington D.C., District of Columbia
  - Howard University College of Medicine, Washington D.C., District of Columbia
  - University of Miami School of Medicine, Miami, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Sinai Hospital of Baltimore Alfred I Coplan Pediatric Hematology Oncology Outpatient Center, Baltimore, Maryland
  - Children's Hospital of Michigan/Wayne State University, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Downstate Medical Center, Brooklyn, New York
  - Duke University Medical Center, Durham, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active | Passive
Started | 130 | 20
Completed | 125 | 18
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Active: Blood and urine specimens, and questionnaires related to the child's health status.
  * Liver Spleen Scan
  * Abdominal Ultrasound
  * Brain magnetic resonance imaging (MRI) / magnetic resonance angiography (MRA)
  * Cardiac Echocardiogram/Pulmonary Function Testing
  * Transcranial Doppler
  * Neuropsychology Testing (Vineland, Wechsler Intelligence Scale for Children (WISC-IV), Connor Continuous Performance Test 2nd Edition (CPT II) and Pediatric Quality of Life Inventory(PedsQOL))
  Patients could be on or off hydroxyurea at the start of Follow-Up Study II, and could change treatment during the study.
- Passive: Information from usual clinical care of sickle cell disease. We will collect information from routine tests ordered by the child's clinical sickle cell doctors.
  Patients could be on or off hydroxyurea at the start of Follow-Up Study II, and could change treatment during the study.
- Total: Total of all reporting groups
Arm/Group | Active | Passive | Total
Number analyzed (Participants) | 130 | 20 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 130 | 20 | 150
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.16 (1.13) | 8.06 (1.26) | 8.15 (1.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 14 | 84
  Male | 60 | 6 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 125 | 19 | 144
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 122 | 18 | 140
  White | 0 | 0 | 0
  More than one race | 4 | 0 | 4
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 130 | 20 | 150

OUTCOME MEASURES:

1. Primary Outcome: Change in Qualitative Spleen Function From Randomized Control Trial Baseline Measurement - Compared Between Children Randomized to Hydroxyurea vs Placebo
Description: The change in splenic function from the randomized control trial baseline measurement was one of the primary outcomes. The change in splenic function (worse vs not-worse) was compared between the randomized treatment groups (hydroxyurea vs placebo). The change in splenic function from baseline (before treatment initiation) to age 10 years (a visit when child turned 10 years old) was defined as worse if it changed from normal to decreased or absent, or decreased to absent; and not worse if it changed from decreased to decreased, normal to normal, decreased to normal, absent to absent, or absent to decreased.
Time Frame: baseline and when child turned 10 years old
Population: All subjects who had age 10 years and baseline spleen function measurement.
Measure: Count of Participants; unit: Participants
Groups:
- Randomized to Hydroxyurea: Subjects randomized to Hydroxyurea in the randomized phase III clinical trial.
- Randomized to Placebo: Subjects randomized to Placebo in the randomized phase III clinical trial.
Arm/Group | Randomized to Hydroxyurea | Randomized to Placebo
Number analyzed (Participants) | 58 | 50
Participants
  Splenic function - worse from baseline | 26 | 28
  Splenic function - not worse from baseline | 32 | 22
Statistical Analysis 1: Comparison: Randomized to Hydroxyurea vs Randomized to Placebo; The primary analysis compared the frequency of worsening spleen function (from normal to decreased or absent, or from decreased to absent); Test type: Superiority; p = 0.33, Fisher Exact

2. Primary Outcome: Change in Qualitative Spleen Function From Randomized Control Trial Baseline Measurement - Compared Between Children on Hydroxyurea vs Off Hydroxyurea at Study Visit
Description: The change in splenic function from the randomized control trial baseline measurement was one of the primary outcomes. The change in splenic function (worse vs not-worse) was compared between children who were known to be on hydroxyurea vs. off hydroxyurea at the time of the visit. The change in splenic function from baseline (before treatment initiation) to age 10 years (a visit when child turned 10 years old) was defined as worse if it changed from normal to decreased or absent, or decreased to absent; and not worse if it changed from decreased to decreased, normal to normal, decreased to normal, absent to absent, or absent to decreased.
Time Frame: baseline and when child turned 10 years old
Population: All subjects who were known to be on hydroxyurea vs. off hydroxyurea at age 10 years, and had age 10 years and baseline spleen function measurement.
Measure: Count of Participants; unit: Participants
Groups:
- On Hydroxyurea at the Time of Visit: Subjects who were on hydroxyurea at the time of study visit
- Off Hydroxyurea at the Time of Visit: Subjects who were off hydroxyurea at the time of study visit
Arm/Group | On Hydroxyurea at the Time of Visit | Off Hydroxyurea at the Time of Visit
Number analyzed (Participants) | 88 | 17
Participants
  Splenic function - worse from baseline | 43 | 9
  Splenic function - not worse from baseline | 45 | 8
Statistical Analysis 1: Comparison: On Hydroxyurea at the Time of Visit vs Off Hydroxyurea at the Time of Visit; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.80, Fisher Exact

3. Primary Outcome: Change in the Percentage of Pitted Cell From Randomized Control Trial Baseline Measurement - Compared Between Children Randomized to Hydroxyurea vs Placebo
Description: The change in the percentage of pitted cell from randomized control trial baseline measurement was one of the primary outcomes. The change in the percentage of pitted cell was compared between the randomized treatment groups (hydroxyurea vs placebo).
Time Frame: Baseline and End of follow-up II study (up to 13 years from randomization date)
Population: All subjects who had end of study and baseline pitted cell measurement.
Measure: Median (Inter-Quartile Range); unit: Percentage of pitted cell
Arm/Group | Randomized to Hydroxyurea | Randomized to Placebo
Number analyzed (Participants) | 70 | 68
Percentage of pitted cell | -1.60 [-5.00 to -0.60] | -1.75 [-6.25 to -0.40]
Statistical Analysis 1: Comparison: Randomized to Hydroxyurea vs Randomized to Placebo; Kruskal-Wallis test was used to test if there were a statistically significant difference between the two treatment groups; Test type: Superiority; p = 0.87, Kruskal-Wallis

4. Primary Outcome: Change in the Percentage of Pitted Cell From Randomized Control Trial Baseline Measurement - Compared Between Children on Hydroxyurea vs Off Hydroxyurea at Study Visit
Description: The change in the percentage of pitted cell from the randomized control trial baseline measurement was one of the primary outcomes. The change in the percentage of pitted cell was compared between children who were known to be on hydroxyurea vs. off hydroxyurea at the time of the visit.
Time Frame: Baseline and End of follow-up II study (up to 13 years from randomization date)
Population: All subjects who were known to be on hydroxyurea vs. off hydroxyurea at the end of study visit, and had end of study and baseline pitted cell count measurement.
Measure: Median (Inter-Quartile Range); unit: Percentage of pitted cell
Arm/Group | On Hydroxyurea at the Time of Visit | Off Hydroxyurea at the Time of Visit
Number analyzed (Participants) | 116 | 22
Percentage of pitted cell | -1.80 [-6.40 to -0.40] | -0.80 [-5.00 to -0.30]
Statistical Analysis 1: Comparison: On Hydroxyurea at the Time of Visit vs Off Hydroxyurea at the Time of Visit; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.28, Kruskal-Wallis

5. Primary Outcome: Change in Howell Jolly Body (HJB) From Randomized Control Trial Baseline Measurement - Compared Between Children Randomized to Hydroxyurea vs Placebo
Description: The change in Howell Jolly Body from the randomized control trial baseline measurement was one of the primary outcomes. The change in Howell Jolly Body was compared between the randomized treatment groups (hydroxyurea vs placebo).
Time Frame: Baseline and End of follow-up II study (up to 13 years from randomization date)
Population: All subjects who had end of follow-up study II and baseline howell jolly body count measurement.
Measure: Median (Inter-Quartile Range); unit: Number of HJB per 10⁶ red blood cell
Arm/Group | Randomized to Hydroxyurea | Randomized to Placebo
Number analyzed (Participants) | 65 | 62
Number of HJB per 10⁶ red blood cell | 2719.88 [1373.90 to 4080.50] | 2248.55 [908.88 to 3758.11]
Statistical Analysis 1: Comparison: Randomized to Hydroxyurea vs Randomized to Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.31, Kruskal-Wallis

6. Primary Outcome: Change in Howell Jolly Body (HJB) Count From Randomized Control Trial Baseline Measurement - Compared Between Children on Hydroxyurea vs Off Hydroxyurea
Description: The change in Howell Jolly Body count from the randomized control trial baseline measurement was one of the primary outcomes. The change in Howell-Jolly Bodies was compared between children who were known to be on hydroxyurea vs. off hydroxyurea at the time of the visit.
Time Frame: Baseline and End of follow-up II study (up to 13 years from randomization date)
Population: All subjects who were known to be on hydroxyurea vs. off hydroxyurea at the end of study visit, and had end of study and baseline Howell Jolly Body count measurement.
Measure: Median (Inter-Quartile Range); unit: Number of HJB per 10⁶ red blood cell
Arm/Group | On Hydroxyurea at the Time of Visit | Off Hydroxyurea at the Time of Visit
Number analyzed (Participants) | 107 | 20
Number of HJB per 10⁶ red blood cell | 2645.43 [1373.90 to 4010.52] | 1833.73 [326.15 to 2713.72]
Statistical Analysis 1: Comparison: On Hydroxyurea at the Time of Visit vs Off Hydroxyurea at the Time of Visit; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.04, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: The date of consent to follow-up study II (FUS-II) through end of FUS-II, up to 4 years
Description: Serious adverse events (SAEs) were Death, Life-threatening event, Prolonged hospitalization (>7 days), Splenic sequestration crisis, Stroke, transient ischemic attack (TIA), Acute chest syndrome, or intensive care unit (ICU) admissions which occurred during the first 5 days following performance of an active assessment study.
  Major events met the definition of SAE but didn't occur within 5 days following the performance of active assessment. These are included below as if they were SAEs.
Groups:
- Randomized to Hydroxyurea: Subjects randomized to Hydroxyurea in the randomized phase III clinical trial.
  150 subjects (130 in active and 20 in passive follow-up group) consented to follow-up II study. Of the 150 subjects, 77 subjects were randomized to the hydroxyurea treatment group during the randomized phase III clinical trial.
- Randomized to Placebo: Subjects randomized to Placebo in the randomized phase III clinical trial.
  150 subjects (130 in active and 20 in passive follow-up group) consented to follow-up II study. Of the 150 subjects, 73 subjects were randomized to the placebo treatment group during the randomized phase III clinical trial.
Arm/Group | Randomized to Hydroxyurea | Randomized to Placebo
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/73
Serious Adverse Events (participants affected / at risk) | 24/77 | 31/73
Other Adverse Events (participants affected / at risk) | 0/77 | 0/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized to Hydroxyurea (N=77) | Randomized to Placebo (N=73)
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 16 (23) | 22 (36)
Vaso-occlusive crisis (Blood and lymphatic system disorders) | 2 (4) | 3 (3)
VOC. Acute hematogenous Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Stroke, TIA (Nervous system disorders) | 1 (1) | 1 (1)
Binocular diplopia and new onset left esotropia (Eye disorders) | 1 (1) | 0 (0)
Pain Crisis (Blood and lymphatic system disorders) | 4 (7) | 5 (6)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Splenic sequestration crisis (Blood and lymphatic system disorders) | 1 (2) | 1 (3)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Bilateral infiltrates on chest x-ray. (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sickle cell anemia with crisis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute hepatic crisis with component of hepatic sequestration. (Hepatobiliary disorders) | 1 (1) | 0 (0)
Delayed hemolytic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lymphangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Osteomyelitis radial (Infections and infestations) | 1 (1) | 0 (0)
Tonsilitis (Infections and infestations) | 0 (0) | 1 (1)
Fever rhinovirus (Infections and infestations) | 1 (1) | 0 (0)
Fever, cough, runny nose, sore throat and difficulty breathing. (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aplastic crisis (Blood and lymphatic system disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Most children used hydroxyurea (HU) for at least part of the FUS-II observation period. This may dilute any effect of randomized group.

Most children were on HU at the specified time points, which reduces power to compare on/off HU.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2006-10-16): https://cdn.clinicaltrials.gov/large-docs/90/NCT01783990/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2009-08-09): https://cdn.clinicaltrials.gov/large-docs/90/NCT01783990/Prot_SAP_001.pdf